CLINICAL TRIAL: NCT00716352
Title: Prospective Registry of Outcomes and Management of Acute Ischaemic Syndromes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Collaborators: Sanofi (Industry); Bristol-Myers Squibb (Industry)
Allocation: Randomized | Model: Parallel | Purpose: Health Services Research
Other Study IDs: MREC/03/10/48
Record Dates: First submitted 2008-07-15; First posted 2008-07-16 (Estimated); Last update posted 2008-07-16 (Estimated); Status verified 2008-07

CONDITIONS: Acute Coronary Syndromes; Coronary Artery Disease
Keywords: non-ST elevation acute coronary syndrome; educational intervention; evidence based practice; guidelines
MeSH Terms: conditions — Acute Coronary Syndrome; Coronary Artery Disease

INTERVENTIONS:
Behavioral: Educational intervention programme

SUMMARY:
This is a multi-centre UK study designed to evaluate if an educational intervention programme delivered to health care professionals can improve the use of evidence based treatments in the management of patients admitted to hospital with non-ST elevation Acute Coronary Syndrome. A total of 38 centres participated, half received the educational intervention. Patients were followed to hospital discharge. Patients were followed up at 6 months. Longer term follow up through the Office Of National Statistics will be performed.

DETAILED DESCRIPTION:
This is a multi-centre UK study designed to evaluate if an educational intervention programme delivered to health care professionals can improve the use of evidence based treatments in the management of patients admitted to hospital with non-ST elevation Acute Coronary Syndrome. A total of 38 centres participated. A cluster randomised method was used and half of centres received the educational intervention. Patients were followed to hospital discharge. Patients were followed up at 6 months and longer term follow up for mortality will be performed through the national databases.

ELIGIBILITY:
Inclusion Criteria:All patients admitted to the hospital (either through casualty or directly to the wards), with a good clinical history of an acute coronary syndrome with one or more of the following:

1. Ischaemic changes on the admission ECG (including patients with bundle branch block)
2. Elevated Troponin or cardiac enzymes on admission
3. Normal ECGs but with evidence of pre-existing coronary artery disease i.e., evidence of a prior history of MI, coronary revascularisation, coronary angiography demonstrating the presence of significant coronary stenosis or a stress test demonstrating ischaemia (treadmill, echo or nuclear scan)

Written informed consent

Exclusion Criteria:

1. Patients with persistent ST elevation >1mm in two or more contiguous leads on the ECG.
2. Patients treated with thrombolytic therapy, or for whom thrombolytic therapy was considered on admission.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1340 (Actual)
Dates: Start 2004-03; Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Adherence to the educational programme measured by the frequency of use of the evidence based treatments: Aspirin, Heparin, Clopidogrel, Beta blockers, Statins.

SECONDARY OUTCOMES:
Comparison of investigations and tests
Use of other treatments
Counselling for lifestyle changes
Referral to smoking cessation clinics
Cardiac rehabilitation
Compliance to treatment at 6 months
Comparison of clinical events at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Flather, Principal Investigator — Royal Brompton & Harefield NHS Trust, Imperial College London
Locations (37):
- United Kingdom (37):
  - University Hospital Aintree, Aintree
  - Monklands Hospital, Airdrie
  - Antrim Hospital, Antrim
  - Barnet General Hospital, Barnet
  - Barnsley District General Hospital, Barnsley
  - Basildon Hospital, Basildon
  - North Hampshire Hospital, Basingstoke
  - Mater Infirmorum Hospital, Belfast
  - Royal Victoria Hospital, Belfast
  - Birmingham Heartlands Hospital, Birmingham
  - Bridlington And District Hospital, Bridlington
  - The Royal Sussex County Hospital, Brighton
  - Cumberland Infirmary, Carlisle
  - Leighton Hospital, Crewe
  - Darent Valley Hospital, Dartford
  - Eastbourne District General Hospital, Eastbourne
  - Western Infirmary, Glasgow
  - Withybush General Hospital, Haverfordwest
  - Altnagelvin Area Hospital, Londonderry
  - Luton and Dunstable Hospital, Luton
  - Macclesfield District General Hospital, Macclesfield
  - Northampton General Hospital, Northampton
  - Royal Alexandra Hospital, Paisley
  - Pontefract General Infirmary, Pontefract
  - Whiston Hospital, Prescot
  - Oldchurch Hospital, Romford
  - Rotherham District General Hospital, Rotherham
  - Hope Hospital, Salford
  - University Hospital Of North Tees, Stockton-on-Tees
  - University Hospital Of North Staffordshire, Stoke-on-Trent
  - Wordsley Hospital, Stourbridge
  - Taunton and Somerset Hospital, Taunton
  - Torbay Hospital, Torquay
  - Pinderfields General Hospital, Wakefield
  - West Cumberland Hospital, Whitehaven
  - Royal Albert Edward Infirmary, Wigan
  - Wrexham Maelor Hospital, Wrexham

REFERENCES:
- See also: Central co-ordinating centre website — http://www.cteu.org